CLINICAL TRIAL: NCT06871722
Title: Effect of Plant-based Diet on Blood Pressure and Gut Microbiota in Kidney Transplant Recipients
Brief Title: How a Plant-Based Diet Affects Blood Pressure and Gut Health in Kidney Transplant Patient
Acronym: PLANET-KT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ramathibodi Ethic ID 6768
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Gut -Microbiota; Kidney Function; Quality of Life (QOL)
Keywords: Plant-based diet; kidney transplant recipient
MeSH Terms: conditions — Hypertension | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: This is a single-center, single-blinded, 1:1 parallel randomized controlled trial. The plant-based diet in this study is defined as a predominantly vegetarian dietary pattern, consisting of two vegetarian meals per day and one meal that includes animal-derived protein. The diet is based on whole foods while avoiding ultra-processed foods.
  Macronutrient Composition Caloric Intake: 30-35 kcal per kilogram of body weight per day Protein Intake: 0.8-1 g per kilogram of body weight per day Fat Sources Animal-derived fats are to be avoided. Plant-based oils are recommended as the primary source of dietary fats. Protein Sources Emphasis is placed on plant-based protein sources, including nuts, beans, edamame, tofu, and tempeh.
  Dairy consumption is permitted, but cow's milk is discouraged. Instead, plant-based alternatives such as almond milk and soy-based milk (e.g., tofu milk) are recommended.
  Egg consumption is allowed but limited to no more than one egg per day
Who Masked: Outcomes Assessor
Masking Description: A biostatistician will generate a random group assignment for participants and inform a research coordinator at the time of randomization. The research coordinator will then inform a RDN each patient's group assignment. Due to the nature of this study, only outcome assessors will be masked; while, patients, the biostatistician, a research coordinator, physicians, and a RDN will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The normal diet for the control group is defined as a standard dietary intake without specific restrictions on protein sources. The dietary guidelines are as follows:
  Caloric Intake: 30-35 kcal per kilogram of body weight per day. Protein Intake: 0.8-1 g per kilogram of body weight per day, with no restrictions on the source of protein.
  Sodium Intake: Participants are encouraged to follow a low-sodium diet, limiting sodium intake to less than 2 g per day, in accordance with dietary recommendations for patients with chronic kidney disease (CKD).
- Plant based diet (Experimental): The plant-based diet in this study is defined as a predominantly vegetarian dietary pattern, consisting of two vegetarian meals per day and one meal that includes animal-derived protein. The diet is based on whole foods while avoiding ultra-processed foods.
  Macronutrient Composition Caloric Intake: 30-35 kcal per kilogram of body weight per day Protein Intake: 0.8-1 g per kilogram of body weight per day Fat Sources Animal-derived fats are to be avoided. Plant-based oils are recommended as the primary source of dietary fats. Protein Sources Emphasis is placed on plant-based protein sources, including nuts, beans, edamame, tofu, and tempeh.
  Dairy consumption is permitted, but cow's milk is discouraged. Instead, plant-based alternatives such as almond milk and soy-based milk (e.g., tofu milk) are recommended.
  Egg consumption is allowed but limited to no more than one egg per day
  Interventions: Behavioral: Plant based diet

INTERVENTIONS:
Behavioral: Plant based diet — The plant-based diet in this study is defined as a predominantly vegetarian dietary pattern, consisting of two vegetarian meals per day and one meal that includes animal-derived protein. The diet is based on whole foods while avoiding ultra-processed foods.
  Macronutrient Composition Caloric Intake: 30-35 kcal per kilogram of body weight per day Protein Intake: 0.8-1 g per kilogram of body weight per day Fat Sources Animal-derived fats are to be avoided. Plant-based oils are recommended as the primary source of dietary fats. Protein Sources Emphasis is placed on plant-based protein sources, including nuts, beans, edamame, tofu, and tempeh.
  Dairy consumption is permitted, but cow's milk is discouraged. Instead, plant-based alternatives such as almond milk and soy-based milk (e.g., tofu milk) are recommended.
  Egg consumption is allowed but limited to no more than one egg per day
  Arms: Plant based diet

SUMMARY:
Kidney transplant improves the quality of life (QoL) and survival of appropriate patients with advanced chronic kidney disease (CKD) and end-stage kidney disease (ESKD). However, these patients still have higher mortality compared to the general population and cardiovascular disease (CVD) is the leading cause of mortality. Among several metabolic complications post-transplantation, hypertension is one of the common risk factors for CVD. In addition to cardiometabolic alteration post-transplant, there is often observed gut microbial dysbiosis, marked by a decrease in microbial diversity and an increase in the relative abundance of Proteobacteria compared to individuals in a healthy state. Different dietary patterns can lead to distinct gut microbiota compositions. Diets rich in plant-based foods, whole grains, fruits, and vegetables tend to promote a more diverse and beneficial gut microbiota characterized by a higher abundance of fiber-degrading bacteria. On the other hand, diets high in saturated fats, refined sugars, and processed foods have been associated with dysbiosis, characterized by a reduction in beneficial bacteria and an overgrowth of potentially harmful microbes. While there is data in the normal population suggesting that a healthy diet can alter gut microbiota composition, the impact of a plant-based diet on gut microbiota-associated hypertension in kidney transplant recipients remains understudied.

To address this gap, the investigators propose a single-center, single-blinded, 1:1 parallel randomized controlled trial to examine the effect of consuming a plant-based diet (intervention group) for 12 weeks on the change in blood pressure, gut microbiota, and patient report outcomes compared to the habitual diet (control group) in kidney transplant recipients with stable kidney allograft function at least 6 months post-transplantation.

The investigators hypothesize that the adoption of a plant-based diet decreases in blood pressure, induces significant changes in gut microbiota composition and does not change in QoL.

DETAILED DESCRIPTION:
Kidney transplantation is the best therapeutic option for patients with advanced CKD and ESKD. It significantly improves quality of life and survival. However, kidney transplant recipients remain facing higher mortality compared to the general population. Similar to the non-transplant population, cardiovascular disease (CVD) is the most common cause of mortality in kidney transplant recipients and hypertension is one of the most common risk factors for CVD. While a plant-based diet is associated with improved blood pressure control, there is a lack of evidence of the benefit of a plant-based diet in kidney transplant recipients. Recently, the gut microbiota has emerged, and the impact appears to be bidirectional. Gut microbiota participates in various effects in the human body such as the synthesis of vitamins, production of short-chain fatty acids, degradation of plant polysaccharides, and immune system development. In CKD, there is alteration in gut microbiota most notably as decrease in the Lactobacillaceae and Prevotellaceae families. After successful kidney transplantation, gut microbial dysbiosis has also been observed and typically characterized by a decrease in microbial diversity and an increase in the relative prevalence of Proteobacteria in comparison to individuals with normal health. Evidence has demonstrated the association of gut microbiota on kidney transplant outcomes such as hypertension, allograft rejection, immunosuppressant metabolism, and post-transplant infection. Therefore, dietary intervention is one of the non-pharmacologic options that can modify and change gut microbiota.

Several types of plant-based diets are associated with beneficial effects on kidney transplant outcomes. For instance, Mediterranean diet is associated with a lower incidence of metabolic syndrome. Dietary Approaches to Stop Hypertension (DASH) diet is associated with a lower risk of kidney allograft function decline and all-cause mortality. Studies have shown the interaction among plant-based dietary consumption, gut microbiota composition, and blood pressure. Although these dietary patterns-related clinical outcomes are associated with improved gut microbiota in kidney transplant recipients, there is a lack of data about the association between consuming plant-based diet, change in gut microbiota, and blood pressure control in kidney transplant recipients. Therefore, the investigators hypothesize that plant-based diet consumption improves blood pressure control and gut microbiota; while, does not decrease the quality of life in kidney transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Receive kidney transplantation after 6 months and before 18 months with a stable kidney allograft function defined by ≤ 25% change in an estimated glomerular filtration rate (eGFR) from the baseline eGFR at 3-month post-transplant for 2 consecutive values closest to the date of randomization. The most recent eGFR before randomization ≥ 30 ml/min/1.73 m2.
* An average SBP ≥ 130 and ≤ 160 mmHg at the time of randomization.
* No change in type and dose of antihypertensive medications ≥ 1 month before randomization or no initiation of new antihypertensive medication ≥ 1 month before randomization
* Anticipated to have no change in type and dose of antihypertensive medications during the 12-week study period.
* Can come to follow up per study protocol.

Exclusion Criteria:

* Combined solid organ transplantation
* Serum sodium < 135 mmol/L before randomization
* Serum potassium > 5.5 mmol/L before randomization
* History of acute kidney allograft rejection of the current kidney allograft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-11-26 (Estimated); Study Completion 2025-11-26 (Estimated)

PRIMARY OUTCOMES:
Difference change of blood pressure | 12 weeks
  The difference in mean blood pressure change at 12 weeks from the baseline between the intervention and control groups.

SECONDARY OUTCOMES:
Gutmicrobiota | 12 weeks
  The difference in gut microbiota composition between the two groups at 12 weeks from baseline, as determined by 16S rDNA sequencing from stool and 3 parameters including alpha diversity, beta diversity, and gut bacterial profile and composition will be evaluated.
Kidney allograft function | 12 weeks
  Change in kidney allograft function between the intervention and control groups, assessed using serum creatinine.
Quality of life by 5EQ-5D-5L score | 12 weeks
  Change in quality of life assessed by 5EQ-5D-5L between intervention and control groups
Kidney allograft function | 12 weeks
  Change in kidney allograft function between the intervention and control groups, assessed using eGFR.

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi Hospial, 270 Rama VI Rd. Thung Phaya Thai, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared. This decision is made to protect participant confidentiality and ensure compliance with institutional and ethical guidelines regarding data privacy